CLINICAL TRIAL: NCT02583217
Title: Effect of Ketamine+Propofol vs Remifentanyl+Propofol on Laryngeal Mask Insertion Conditions
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, MD, Ankara University
Other Study IDs: ANK-42476
Record Dates: First submitted 2015-09-18; First posted 2015-10-22 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2016-01

CONDITIONS: Surgery
Keywords: Laryngeal mask; Ketamine; Remifentanyl
MeSH Terms: interventions — Ketamine; Remifentanil; Propofol; Laryngeal Masks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ketamine: Ketamine+propofol
  Interventions: Drug: Ketamine; Drug: propofol; Device: laryngeal mask
- Remifentanyl: Remifentanyl+propofol
  Interventions: Drug: remifentanyl; Drug: propofol; Device: laryngeal mask

INTERVENTIONS:
Drug: Ketamine — To compare ketamine+propofol versus remifentanyl+propofol to maintain good laryngeal mask insertion conditions
  Other Names: Remifentanyl
  Groups: Ketamine
Drug: remifentanyl
  Groups: Remifentanyl
Drug: propofol
Device: laryngeal mask

SUMMARY:
Laryngeal mask airway is a common tool for airway management during anesthesia in many surgeries. Insertion of laryngeal mask needs deep anesthesia, suppression of airway, stabile hemodynamic response. Many drug regimens has been used for this purpose. This study aimed to compare the insertion conditions of laryngeal mask by using ketamine+propofol versus remifentanil + propofol.

ELIGIBILITY:
Inclusion Criteria:

* Surgery requires laryngeal mask

Exclusion Criteria:

* Patient refusal, abdominal surgery required muscle relaxant, any allergy to ketamine or remifentanyl

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgery performed with laryngeal mask as airway tool in gynecologic clinic
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
High laryngeal mask insertion scores | 3 minutes

SECONDARY OUTCOMES:
Hypotension | 10 minutes
Hypertension | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIM GUCLU, MD, Principal Investigator — Ankara University
Locations (1):
- Cigdem Yildirim Guclu, Ankara, Turkey (Türkiye)